CLINICAL TRIAL: NCT04507126
Title: Effects of Bacillus Calmette-Guérin (BCG) Immunization on Cerebrospinal Fluid (CSF) and Blood-Based Biomarkers in Older Adults: A Pilot
Brief Title: A Pilot Study of the Effects of BCG Immunization on CSF and Blood-based Biomarkers in Older Adults.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven E Arnold, MD, Professor of Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020P002042; 2021P001980 (Other: MGB IRB)
Record Dates: First submitted 2020-06-23; First posted 2020-08-11 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Cognition; Alzheimer's disease; Memory; BCG; Immunization
MeSH Terms: conditions — Alzheimer Disease | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCG Immunization (Experimental): All participants will receive two Bacillus Calmette-Guérin (Japan BCG) vaccine injections spaced four week apart. Each injection will have 1.8-3.9 x 10^6 colony forming units (CFU) reconstituted in 0.1 mL saline.
  Interventions: Biological: Bacillus Calmette-Guerin (BCG)

INTERVENTIONS:
Biological: Bacillus Calmette-Guerin (BCG) — Vaccine

SUMMARY:
A pilot study of the effects of Bacillus Calmette-Guérin (BCG) immunization on cerebrospinal fluid and blood-based biomarkers in older adults.

DETAILED DESCRIPTION:
This single-site, open-label clinical trial will investigate the immune and neurobiological effects of BCG vaccination in cognitively unimpaired older adults and older adults with memory and thinking problems by measuring target engagement, pharmacodynamic response, and effect on Alzheimer's disease (AD) pathology and immune response markers. This study will also gather data on study feasibility, tolerability, and safety.

ELIGIBILITY:
Inclusion Criteria:

Study subjects meeting all the following criteria will be allowed to enroll in the study:

1. Age 55-80 inclusive;
2. Montreal Cognitive Assessment (MoCA ) ≥18;
3. Normal cognition as defined by Montreal Cognitive Assessment (MoCA) ≥ 26 or Mild Cognitive Impairment (MCI) as defined by the National Institute of Health Alzheimer's Association (NIA-AA) Workgroup (2011) and MoCA score between 18 and 25 (inclusive);
4. Education level, English language skills, and literacy indicates subject will be able to complete all assessments;
5. Ability to provide informed consent;
6. Willing and able to complete all assessment and study procedures, including blood draws, lumbar punctures, and clinical assessments;
7. If on cholinesterase inhibitor and/or memantine, doses are stable for 3 months prior to baseline;
8. Negative test results for Human Immunodeficiency Virus (HIV) antibody and Tuberculosis (TB) (QuantiFERON) at screening;
9. No prior Bacillus Calmette-Guérin (BCG) exposure either through birth vaccinations (born in North American) or BCG bladder cancer treatment.
10. Documentation of current flu season vaccination dated at least 60 days prior to baseline visit.

Exclusion Criteria:

Study subjects meeting any of the following criteria will not be allowed to enroll in the study:

1. History of chronic infectious disease, such as HIV or untreated or active hepatitis;
2. History of tuberculosis, positive interferon-gamma release assay (IGRA, also known as the QuantiFERON-TB test), including a test with a high reactivity to mycobacteria of non-tuberculosis variety;
3. Prior BCG vaccination, positive T-spot tuberculosis test or a T-spot test showing significant Mycobacteria exposure;
4. A positive Severe acute respiratory syndrome coronavirus, Polymerase Chain Reaction (PCR) result within 3 months of screening, or known close contact with a confirmed Coronavirus 19 (COVID-19) positive person or symptoms highly suspicious for COVID-19 (per Center for Disease Control (CDC) guidelines) within 1 month of screening, including fever, cough, shortness of breath, chills, muscle pain, new loss of taste or smell, vomiting or diarrhea, and/or sore throat, based on clinician's judgment;
5. History of treatment with metformin within the past one year;
6. Previous participation (ever) in active immunization research for Alzheimer's Disease (AD) or passive immunotherapy or other disease-modifying treatments for AD within the past three months;
7. Current treatment with immunosuppressants (calcineurin inhibitors, corticosteroids, or biological or cytotoxic immunosuppressants, or disease or condition likely to require high dose steroid or immunosuppressive therapy);
8. Other conditions or treatments associated with increased risk of infections or treatment with immunosuppressive medications for any reason;
9. Current treatment with aspirin > 160 mg/day or chronic, daily nonsteroidal anti-inflammatory drugs (NSAIDs);
10. Chronic use of antibiotics;
11. History of keloid formation;
12. Living with someone who is immunosuppressed and/or at high risk for infectious diseases (for example, HIV+ or taking immunosuppressive medications for any reason), or in a job (e.g. healthcare) in which the subject works with immunosuppressed populations;
13. Other/confounding neurological or psychiatric condition, unstable medical or psychiatric conditions, contraindications to BCG use and lab abnormalities or concurrent medication use posing risk for BCG or study procedures;
14. Laboratory abnormalities in B12, Folate, thyroid stimulating hormone (TSH), or other common laboratory parameters that may contribute to cognitive dysfunction;
15. Laboratory abnormalities in Complete Blood Count (CBC), electrolytes, Liver Function Tests (LFTs), Blood Urea Nitrogen (BUN), Creatinine (Cr), total serum immunoglobulins, erythrocyte sedimentation rate (ESR), C reactive protein (CRP), or urinalysis posing risk to treatment with BCG per clinician judgment;
16. Laboratory abnormalities in prothrombin time /international normalized ratio (PT-INR), which would pose a risk to performing the lumbar puncture procedure;
17. Discontinuation of cholinesterase inhibitor or memantine within one month (28 days) prior to baseline visit;
18. Females who are pregnant, lactating or of child-bearing potential;
19. If male with female partner(s) of childbearing potential, unwilling or unable to adhere to contraception requirements specified in the protocol.
20. Administration of live vaccine <60 days prior to Baseline.
21. Increased intracranial pressure as determined on a fundoscopy/neurological examination performed within 30 days of Lumbar Puncture (LP);
22. COVID-19 vaccination < 60 days prior to baseline or within 14 days of BCG immunizations.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Arnold, MD, Principal Investigator — Massachusetts General Hospital; Denise Faustman, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical Translational Research Unit, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCG Immunization
Started | 20
Enrolled | 20
Completed | 13
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | BCG Immunization
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  55-80 Years Old | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - caucasian/european heritage | 16
  Non Hispanic | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Cerebrospinal Fluid (CSF) collection [Count of Participants; unit: Participants] | 16
Blood collection [Count of Participants; unit: Participants] | 16
Number of participants that participated in cognitive testing [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: Median Fold Change of Cytokine Levels From Day 0 to Day 90
Description: Heat-killed BCG or Lipopolysaccharide (LPS) applied to peripheral blood mononuclear cells (PBMCs) from subjects at 0 and 90d after study start.
  Calculated as median fold change of cytokine levels in media at day 90 (pg/mL) compared to day 0 (pg/mL)
Time Frame: Day 90 compared to Day 0
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | BCG Immunization
Number analyzed (Participants) | 10
pg/mL
  Interferon-gamma cytokine | 3254 [281.1 to 7169]
  Interleukin-1 beta cytokine | 1.997 [-5.641 to 15.08]
  Interleukin 6 cytokine | 16.83 [-319.8 to 717.5]
  Tumor necrosis factor alpha cytokine | -33.89 [-529.3 to 1746]

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Number of Participants With Treatment-Related Adverse Events to determine safety of BCG
Time Frame: AEs were collected from baseline through study completion, an average of 390 days
Measure: Count of Participants; unit: Participants
Groups:
- BCG Immunization: All participants will receive two Bacillus Calmette-Guérin (Japan BCG) vaccine injections spaced four week apart. Each injection will have 1.8-3.9 x 10^6 colony forming units (CFU) reconstituted in 0.1 mL saline.
  Number of Participants With Treatment-Related Adverse Events to determine safety of BCG
Arm/Group | BCG Immunization
Number analyzed (Participants) | 16
Participants | 0

3. Secondary Outcome: Median Difference in CSF Biomarkers of Alzheimer's Disease (AD) Pathology From Day 0 to Day 90
Description: Median difference of biomarkers measured in pg/mL (Amyloid-β42/40, phospho-tau (p181 tau), glial fibrillary astrocytic protein (GFAP) and neurofilament light protein (NFL) biomarkers) in CSF from baseline to 90 days.
Time Frame: Day 90 compared to Day 0
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | BCG Immunization
Number analyzed (Participants) | 15
pg/mL
  AB42/40 | -0.0005220 [-0.002264 to 0.002382]
  NFL | -47.17 [-361.6 to 125.7]
  GFAP | 789.7 [-693 to 3842]
  p181- Tau | 1.058 [-.9333 to 4.767]

4. Secondary Outcome: Median Fold Change in CSF Biomarkers of Pharmacodynamic Response From Day 0 to Day 90
Description: Median Fold change in CSF biomarkers from baseline measured in pg/mL (Interleukin 6 (IL6), Tumor Necrosis Factor alpha (TNFa), interleukin 1 beta (IL1beta), Interferon gamma (IFNg))
Time Frame: Day 90 compared to Day 0
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | BCG Immunization
Number analyzed (Participants) | 16
pg/mL
  Interferon gamma (IFNg) | -.01 [-3.015 to 4.500]
  Interleukin 6 (IL6) | 7.332 [-783 to 548.2]
  Tumor Necrosis Factor alpha (TNFa) | -.8676 [-14.66 to 6.242]
  Interleukin 1 beta (IL1B) | 23.74 [-7.202 to 72.03]

5. Secondary Outcome: Cognitive Measures (RBANS) Total Scored Index, 3 Months After BCG Injection
Description: Mean change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) from baseline to 3 months after BCG injection. Total Scaled Index (TSI) . Higher scores mean better performance on the RBANS Total Scaled Index.
  TSI Minimum 40, TSI Maximum 160.
Time Frame: Day 90 compared to Day 0
Measure: Mean (95% Confidence Interval); unit: units on TSI scale
Arm/Group | BCG Immunization
Number analyzed (Participants) | 16
units on TSI scale
  Day 0 | 98.1 [88.57 to 107.7]
  Day 90 | 104.1 [93.32 to 114.8]

6. Secondary Outcome: Median Fold Change in Circulating Cytokines From Day 0 to Day 90
Description: Median Fold change in circulating cytokines in plasma from baseline measured in pg/mL (IL6, TNFa, IL1beta, IFNg)
Time Frame: Time Frame: Day 90 compared to Day 0
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | BCG Immunization
Number analyzed (Participants) | 16
pg/mL
  IFNg | 259.8 [27.32 to 789.4]
  IL1beta | 33.47 [-20.48 to 109.1]
  IL6 | 332.9 [-769.4 to 1020]
  TNFa | 24.80 [-22.71 to 145.8]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to end of study, up to 396 days.
Description: Adverse events were systematically collected at each study visit and reviewed by the study PI regularly.
Arm/Group | BCG Immunization
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG Immunization (N=16)
Post Lumbar Puncture Headache (Nervous system disorders) | 4 (4)
Intermittent headache (Nervous system disorders) | 2 (2)
Back pain (Nervous system disorders) | 3 (3)
Fatigue (Nervous system disorders) | 2 (2)
Hematoma at blood draw site (Skin and subcutaneous tissue disorders) | 1 (1)
Removal of squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Increased stress (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04507126/Prot_SAP_000.pdf